CLINICAL TRIAL: NCT01307397
Title: An Open-Label, Multicenter Study to Assess the Safety of RO5185426 (Vemurafenib) in Patients With Metastatic Melanoma
Brief Title: A Study of Vemurafenib in Participants With Metastatic Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO25515; 2010-023526-21 (EudraCT Number)
Record Dates: First submitted 2011-02-17; First posted 2011-03-02 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (1):
- Vemurafenib (Experimental): Participants will receive vemurafenib at a dose of 960 milligrams (mg) twice daily (bid) until the development of progressive disease, unacceptable toxicity, consent withdrawal, protocol violations endangering participant's safety, death, or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Participants will receive continuous oral doses of vemurafenib 960 mg (four 240 mg tablets) twice daily in each 28-day treatment cycle until the development of progressive disease, unacceptable toxicity, consent withdrawal, protocol violations endangering participant's safety, death, or study termination by the Sponsor, whichever occurs first.
  Other Names: RO5185426, Zelboraf

SUMMARY:
This multi-center study evaluates the safety and efficacy of vemurafenib in participants with BRAF V600 mutation-positive, surgically incurable, and unresectable Stage IIIC or IV (American Joint Committee on Cancer [AJCC]) metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Histologically confirmed metastatic melanoma (surgically incurable and unresectable Stage IIIC or Stage IV; AJCC) with BRAF V 600 mutation determined by Cobas 4800 BRAF Mutation Test. Unresectable Stage IIIC disease must have had confirmation from a surgical oncologist
* Participants with either measurable or non-measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1
* Participants may or may not have received prior systemic therapy for metastatic melanoma
* Eastern Cooperative Oncology Group (ECOG) performance status between 0 to 2
* Adequate hematologic, renal and liver function

Exclusion Criteria:

* Evidence of symptomatic central nervous system (CNS) lesions, use of steroids or anti-seizure medications for treatment of brain metastases prior to the first administration of vemurafenib
* Previous malignancy (other than melanoma) within the past 2 years, except for treated and controlled basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix
* Concurrent administration of any anti-cancer therapies other than those administered in the study
* Clinically significant cardiovascular disease or event within the 6 months prior to first administration of study drug
* Refractory nausea or vomiting, external biliary shunt, or significant bowel resection that would preclude adequate absorption

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3219 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (280):
- University "Mother Theresa" Hospital Center; Oncology Department, Tirana, Albania
- Argentina (3):
  - Hospital Britanico; Oncologia, Buenos Aires
  - Fundación CIDEA, Buenos Aires
  - Inst. Alexander Fleming; Oncologia, Buenos Aires
- Australia (12):
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Newcastle Mater Misericordiae Hospital; Oncology, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Border Medical Oncology, Wodonga, New South Wales
  - Greenslopes Private Hospital; Gallipoli Research Centre, Greenslopes, Queensland
  - The Townsville Hospital; Townsville Cancer Centre, Townsville, Queensland
  - Princess Alexandra Hospital Woolloongabba; Clinical Hematology and Medical Oncology, Woolloongabba, Queensland
  - Royal Adelaide Hospital; Oncology, Adelaide, South Australia
  - Geelong Hospital; Geelong Cardiology Practice, Geelong, Victoria
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (8):
  - Landeskrankenhaus Feldkirch; Abteilung für Innere Medizin, Feldkirch
  - LKH Graz; Abteilung für allgemeine Dermatologie, Graz
  - LKH Innsbruck; Universitätsklinik für Dermatologie, Innsbruck
  - Krankenhaus der Elisabethinen Linz; Abteilung für Dermatologie, Linz
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - LKH Salzburg; Universitätsklinik für Dermatologie, Salzburg
  - Landesklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien; Univ.Klinik für Dermatologie, Vienna
- Belgium (3):
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - Sint Augustinus Wilrijk, Wilrijk
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Brazil (5):
  - Instituto Nacional de Cancer - INCa; Pesquisa Clinica, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital A. C. Camargo; Oncologia, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- Bulgaria (2):
  - District Oncology Dispensary; Department for Oncology and Dermatology, Plovdiv
  - National Specialized Hospital for Active Oncology Treatment; Dermatology Clinic, Sofia
- Canada (12):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Lion'S Gate Hospital, North Vancouver, British Columbia
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - St. Boniface General Hospital; Medicine, Winnipeg, Manitoba
  - QEII HSC; Oncology, Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - The Ottawa Hospital; Division of Infectious Diseases, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - Chuq - Hopital Hotel Dieu de Quebec; Oncology, Québec, Quebec
- Colombia (4):
  - Centro Javeriano de Oncología, Bogotá
  - Fundacion Santa Fe de Bogotá, Bogotá
  - Clínica Imbanaco; Oncology, Cali
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
- Clinical Hospital Sisters of Mercy, Zagreb, Croatia
- Czechia (6):
  - Masarykův onkologický ústav; Klinika komplexní onkologické péče, Brno
  - University Hospital; Oncology and Radiotherapy, Hradec Králové
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Faculty Hospital; Dialysis Unit, Ostrava
  - 1 Lekarska Fakulta Uni Karlovy; 3 Interni Klinika, Labor. Pro Endokrinologii A Metabolismus, Prague
  - Faculty Hospital Kralovske Vinohrady; Oncology, Prague
- Denmark (3):
  - Aarhus Universitetshospital; Kræftafdelingen, Aarhus C
  - Herlev Hospital; Onkologisk afdeling, Herlev
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense
- Ecuador (3):
  - Hospital Regional Vicente Corral Moscoso, Servicio de Oncología, Cuenca
  - Hospital Abel Gilbert Ponton; Oncology, Guayaquil
  - Hospital Solca Portoviejo; Oncologia, Portoviejo
- Estonia (3):
  - East Tallinn Central Hospital; Clinic of Internal Medicine, Tallinn
  - North Estonia Medical Centre Foundation; Oncology Center, Tallinn
  - Tartu University Hospital; Clinic of Hematology and Oncology, Tartu
- Finland (3):
  - Helsinki University Central Hospital; Dept of Oncology, Helsinki
  - Tampere University Hospital; Dept of Oncology, Tampere
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- Germany (43):
  - Uniklinik RWTH Aachen; Klinik für Dermatologie und Allergologie - Hautklinik, Aachen
  - Klinikum Augsburg Süd; Klinik für Dermatologie und Allergologie, Augsburg
  - CAMPUS BENJAMIN FRANKLIN CharitéCentrum 14 Med.Klinik f.Hämatologie u.Onkologie, Berlin
  - St. Josef-Hospital Klinik f. Dermatologie u. Allergologie, Bochum
  - Elbekliniken Buxtehude; Klinik für Dermatologie, Buxtehude
  - DRK-Krankenhaus; Hautklinik, Chemnitz
  - Klinik der Uni zu Köln; Klinik & Poliklinik fuer Dermatologie & Venerologie, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Düsseldorf; Hautklinik, Düsseldorf
  - HELIOS Klinikum Erfurt, Klinik für Hautkrankheiten und Allergologie, Erfurt
  - Universitätsklinikum Erlangen; Hautklinik, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Klinik fuer Allgemein- und Viszeralchirurgie, Frankfurt
  - Uniklinikum Freiburg Dermatol, Freiburg im Breisgau
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - Universitätsmedizin Göttingen Georg-August-Universität Zentrum Dermatologie, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf Zentrum f.Innere Medizin Klinik f.Dermatologie, Hamburg
  - Medizinische Hochschule; Hautklinik Linden, Hanover
  - Uni-Hautklinik, Heidelberg
  - Klinikum am Gesundbrunnen; Tumorzentrum, Heilbronn
  - Universitätsklinikum Jena; Klinik für Hautkrankheiten, Jena
  - Klinikum Kassel; Hautklinik, Kassel
  - UNI-Klinikum Campus Kiel Klinik f.Dermatologie Tagesklinik f.Dermatologie, Kiel
  - Universitätsklinikum Leipzig Klinik f.Dermatologie Venerologie u.Allergologie, Leipzig
  - Klinikum d.Stadt Ludwigshafen Hautklinik, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein; Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg; Hautklinik; Klinik für Dermatologie und Venerologie, Magdeburg
  - Johannes Gutenberg Unis-Klinik; Dept For Dermatology, Mainz
  - Klinikum Mannheim Klinik fuer Dermatologie, Venerologie und Allergologie, Mannheim
  - Universitätsklinikum Marburg Klinik f. Dermatologie, Marburg
  - Johannes-Wesling-Klinikum Minden; Onkologische Ambulanz / Tagesklinik, Minden
  - Klinikum der LMU München; Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Staedtisches Krankenhaus Muenchen-Schwabing, Haematologie & Onkolgie, München
  - Universitätsklinikum Münster, Münster
  - Fachklinik Hornheide; Internistische Onkologie, Münster
  - Klinikum Nürnberg Nord; Hautklinik; Klinik für Dermatologie, Nuremberg
  - Klinikum Dorothea Ch.Erxleben; Klinik für Dermatologie und Allergologie, Quedlinburg
  - KLINIKUM VEST GmbH Knappschaftskrankenhaus Abt.Haut- Allergie- Venen- und Umwelterkrankungen, Recklinghausen
  - Universitätsklinikum Regensburg; Klinik und Poliklinik für Dermatologie, Regensburg
  - Universitaets-Hautklinik Tuebingen, Tübingen
  - Wilhelm Fresenius Klinik; Klinik f. Dermatologie u. Allergologie, Wiesbaden
  - HELIOS Klinikum Barmen Zentrum Dermatologie Allergologie und Umweltmedizin, Wuppertal
  - Universitätsklinikum Würzburg; Klinik und Poliklinik für Dermatologie Venerologie u. Allergologie, Würzburg
- Greece (4):
  - Laiko General Hospital; 1St Pathological Clinic, Athens
  - Hospital Hygeia; 1St Oncology Dept., Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - Metropolitan Hospital; Dept. of Oncology, Piraeus
- Hungary (5):
  - Semmelweis Egyetem; Bor-, Nemikortani es Boronkologiai Klinika, Budapest
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Debreceni Egyetem OEC; Borgyogyaszati Klinika, Debrecen
  - Pecsi Tudomanyegyetem AOK; Borgyogyaszati Klinika, Pécs
  - Szegedi Tud.Egyetem Szent-Gyorgyi Albert Klin.Kozp., Szeged
- India (7):
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Rajiv Gandhi Cancer Inst.&Research Center; Medical Oncology, New Delhi, National Capital Territory of Delhi
  - Basavatarakam Indo-American Cancer Hospital & Research Institute, Hyderabad
  - Chhatrapati Shahuji Maharaj Medical University; Department of Oncology, Lucknow
  - Regional Cancer Centre; Dept of Oncology, Trivandrum
  - Christian Med Clg & Hspt, Vellore
- Ireland (8):
  - Cork Uni Hospital; Oncology Dept, Cork
  - St Vincent'S Uni Hospital; Medical Oncology, Dublin
  - Mater Misericordiae Uni Hospital; Oncology, Dublin
  - Mater Private Hospital, Dublin
  - St James' Hospital; Cancer Clinical Trials Office, Dublin
  - Galway Uni Hospital; Oncology Dept, Galway
  - University Hospital Limerick - Oncology, Limerick
  - Waterford Regional Hospital; Department Of Medical Oncology, Waterford
- Israel (4):
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Ranbam Health Care Campus; Oncology - Hafia, Hafia
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
- Italy (21):
  - Istituto Tumori Giovanni Paolo II IRCSS; Ospedale Oncologico Bari, Bari, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - AO Santa Maria Nuova; U.O. Day Hospital di Oncologi, Reggio Emilia, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia, Udine, Friuli Venezia Giulia
  - Istituto Dermopatico dell'Immacolata (IDI)-IRCCS; IV Divisione Oncologica e Dermatologia Oncologica, Rome, Lazio
  - IFO - Istituto Regina Elena; Oncologia Medica, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - Az. Osp. Spedali Civili; Divisione Di Oncologia - Iii Medicina, Brescia, Lombardy
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Policlinico Le Molinette; Clinica Dermatologica, Turin, Piedmont
  - Policlinico P. Giaccone; Istituto Di Oncologia, Clinica Medica 1, Palermo, Sicily
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - Azienda Ospedaliera S. Chiara; Dip di Onc,Trapianti e delle Nuove Tecnologie in Medicina, Pisa, Tuscany
  - A.O.U. Senese Policlinico Santa Maria Alle Scotte, Siena, Tuscany
  - Azienda Ospedaliera S. Maria - Terni; Oncologia, Terni, Umbria
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
- Latvia (2):
  - Daugavpils Regional Hospital, Daugavpils
  - Rigas Austrumu Kliniska Universitates slimnica, Latvijas Onkologijas centrs, Riga
- Lithuania (2):
  - Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Hematology, Oncology and Tranfusion Medicine Center, Vilnius
- Mexico (3):
  - Fundación Rodolfo Padilla Padilla, A.C.; Oncology, León
  - Hospital General de México; Unidad de Oncologia, Mexico City
  - Inst. Nacional de Cancerologia; Investigacion Clinica, Mexico City
- Netherlands (10):
  - Antoni Van Leeuwenhoek Ziekenhuis; Inwendige Geneeskunde, Amsterdam
  - VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam
  - Tergooiziekenhuizen, Blaricum
  - Amphia Ziekenhuis, Breda
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Academisch Ziekenhuis Leiden; Clinical Oncology, Leiden
  - Academish Ziekenhuis Maastricht (Azm); Inwendige Geneeskunde, Maastricht
  - UMC St Radboud; Interne Oncologie; Medical Oncology Department, Nijmegen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht; Inwendige Geneeskunde Afd., Utrecht
- University Clinic for Radiotherapy and Oncology Skopje; Department of skin malignancies, Skopje, North Macedonia
- Norway (2):
  - Haukeland Universitetshospital; Onkologisk Avd., Bergen
  - The Norvegian Radium Hospital Montebello; Dept of Oncology, Oslo
- Peru (2):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud; Oncology & Haemathology, Arequipa
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
- Poland (4):
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - ZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii;Wojska Polskiego 37, Olsztyn
  - NZOZ Med.-Polonia sp. z o.o., Poznan
  - Centrum Onkologii- Instytut; im. M.Skłodowskiej-Curie, Warsaw
- Portugal (2):
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Romania (3):
  - Institut of Oncology Al. Trestioreanu Bucharest; Oncology, Bucharest
  - Medisprof SRL, Cluj-Napoca
  - S.C. Life Search S.R.L; Medical Oncology Clinic, Timișoara
- Russia (7):
  - FSBI "Scientific Research Institute of Oncology named after N.N.Petrov" Ministry of Health of RF, Saint Petersburg, Sankt-Peterburg
  - Regional Clinical Oncology Dispensary, Krasnodar
  - Russian Cancer Research Center, Moscow
  - Moscow city oncology hospital #62 of Moscow Healthcare Department, Moscow
  - St. Petersburg Oncology & Gynecology; City Clinical Oncology Dispensary, Saint Petersburg
  - Stavropol Clinical Oncology Dispansary, Stavropol
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Clinical Center Bezanijska Kosa; Oncology, Belgrade
- Slovakia (3):
  - Onkologicky ustav sv. Alzbety; Oddelenie ambulantnej chemoterapie, Bratislava
  - Narodny Onkologicky Ustav; Oddelenie klinickej onkologie E, Bratislava
  - POKO Poprad; Department of Oncology, Poprad
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (6):
  - Universitas Annex, University of the Free State; Clinical Oncology, Bloemfontein
  - Cape Town Oncology Trials, Cape Town
  - Cancercare, Cape Town
  - Medical Oncology Centre of Rosebank; Oncology, Johannesburg
  - Steve Biko Academic Hospital; Oncology, Pretoria
  - Sandton Oncology Centre, Sandton
- South Korea (5):
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Seoul National University Hosp; Dept Internal Med Hem Onc, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Asan Medical Center., Seoul
- Spain (27):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña, La Coruña
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Santa Lucía; Servicio de Oncología Médica, Cartagena (Murcia), Murcia
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Xeral Cíes; Servicio de Oncologia, Vigo, Pontevedra
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias (HUC), La Laguna (Tenerife), Tenerife
  - Hospital de Cruces; Servicio de Oncologia, Barakaldo, Vizcaya
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves; Servicio de Oncologia, Granada
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset; Onkology, Gothenburg
  - Skånes Onkologiska Klinik, Universitetssjukhuset, Lund
  - Karolinska Universitetssjukhuset, Solna, Stockholm
  - Norrlands universitetssjukhus; Onkologkliniken, Umeå
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Switzerland (6):
  - Universitaetsspital Basel; Onkologie, Basel
  - Inselspital Bern; Medizinische Onkologie, Bern
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
  - CHUV; Departement d'Oncologie, Lausanne
  - Kantonsspital St. Gallen; Onkologie/Hämatologie, Sankt Gallen
  - Universitätsspital Zürich; Dermatologische Klinik, Zurich
- Turkey (Türkiye) (12):
  - Adana Baskent University Hospital; Medical Oncology, Adana
  - Cukurova Uni Faculty of Medicine; Medical Oncology, Adana
  - Ankara Uni , Ibn-I Sina Hospital; Oncology Dept, Ankara
  - Gazi Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Akdeniz University School of Medicine; General Surgery, Antalya
  - Ege University Medical Faculty; Medical Oncology Department, Bornova, İ̇zmi̇r
  - Gaziantep University Medical Faculty, Medical Oncology Department, Gaziantep
  - Kartal Training and Research Hospital;Medical Oncology Department, Istanbul
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - American Hospital, Medical Oncology Department, Istanbul
  - Dokuz Eylul Uni ; Medical Oncology, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara
- United Kingdom (12):
  - Addenbrookes Nhs Trust; Oncology Clinical Trials Unit, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital; St. Lukes Cancer Centre, Guildford
  - St James University Hospital, Leeds
  - Royal Marsden Hospital, London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Northern Centre for Cancer Care Freeman Hospital; Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne
  - Mount Vernon Hospital; Centre For Cancer Treatment, Northwood
  - Nottingham University Hospitals City Campus, Nottingham
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Southampton General Hospital; Medical Oncology, Southampton
  - Singleton Hospital; Oncology, Swansea

REFERENCES:
- [Derived] Larkin J, Brown MP, Arance AM, Hauschild A, Queirolo P, Vecchio MD, Ascierto PA, Krajsova I, Schachter J, Neyns B, Garbe C, Sileni VC, Mandala M, Gogas H, Espinosa E, Hospers G, Lorigan P, Nyakas M, Guminski A, Liszkay G, Rutkowski P, Miller W Jr, Donica M, Makrutzki M, Blank C. An open-label, multicentre safety study of vemurafenib in patients with BRAFV600-mutant metastatic melanoma: final analysis and a validated prognostic scoring system. Eur J Cancer. 2019 Jan;107:175-185. doi: 10.1016/j.ejca.2018.11.018. Epub 2018 Dec 20. PMID 30580112
- [Derived] Larkin J, Del Vecchio M, Ascierto PA, Krajsova I, Schachter J, Neyns B, Espinosa E, Garbe C, Sileni VC, Gogas H, Miller WH Jr, Mandala M, Hospers GA, Arance A, Queirolo P, Hauschild A, Brown MP, Mitchell L, Veronese L, Blank CU. Vemurafenib in patients with BRAF(V600) mutated metastatic melanoma: an open-label, multicentre, safety study. Lancet Oncol. 2014 Apr;15(4):436-44. doi: 10.1016/S1470-2045(14)70051-8. Epub 2014 Feb 27. PMID 24582505

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib: Participants received continuous oral doses of vemurafenib 960 milligrams (mg) (four 240 mg tablets) twice daily in each 28-day treatment cycle until the development of progressive disease, unacceptable toxicity, consent withdrawal, protocol violations endangering participant's safety, death or study termination by the Sponsor.
Period: Overall Study
Arm/Group | Vemurafenib
Started | 3219
Completed | 3219 (A participant completed study in case of progressive disease, adverse events or consent withdrawn)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of study medication.
Groups:
- Vemurafenib: Participants received continuous oral doses of vemurafenib 960 mg (four 240 mg tablets) twice daily in each 28-day treatment cycle until the development of progressive disease, unacceptable toxicity, consent withdrawal, protocol violations endangering participant's safety, death or study termination by the Sponsor.
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1397
  Male | 1822

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Grade 3 or 4 Adverse Events (AEs) as Determined by National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 4.0
Description: The intensity of AEs were graded on a 5-point scale (Grade 1 to 5) according to the NCI-CTCAE version 4.0, where Grade 1 indicates "Mild" severity and Grade 5 indicates "Death". The CTCAE defines Grades 3 and 4 as follows: Grade 3 means "Severe"; Inability to work or perform normal daily activity; treatment or medical intervention is indicated in order to improve the overall well-being or symptoms; delaying the onset of treatment is not putting the survival of the participant at direct risk. Grade 4 means "Life-threatening, Disabling"; based on extreme limitation in activity; significant medical intervention/therapy required; and hospitalization probable.
Time Frame: Baseline up to 28 days post end of treatment (maximum up to 46 months)
Population: Safety population. Number of participants analyzed = participants with measurable disease at baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of participants | 52.8

2. Primary Outcome: Percentage of Participants With at Least 1 AE Leading to Study Drug Interruption or Drug Discontinuation
Description: An AE was considered as any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Pre existing conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. Percentage of participants with dose interruption or discontinuation due to AE was presented.
Time Frame: Baseline up to 28 days post end of treatment (maximum up to 46 months)
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of participants
  AE Leading to Drug Discontinuation | 7.0
  AE Leading to Study Drug Interruption | 34.0

3. Primary Outcome: Percentage of Participants With AEs of Special Interest
Description: AEs of special interest included cutaneous squamous cell carcinoma (SCC), rash, photosensitivity, liver injury, arthralgia, fatigue, gastrointestinal (GI) polyps, pancreatitis, potentiation of radiation toxicity, prolongation of cardiac repolarization or arrhythmia, non-cutaneous SCC and other primary malignancies (other than cutaneous SCC or new primary melanoma).
Time Frame: Baseline up to 28 days post end of treatment (maximum up to 46 months)
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of participants
  Arthralgia | 42.3
  Rash | 47.9
  Photosensitivity | 28.4
  Fatigue | 36.8
  Cutaneous SCC | 14.6
  Non Cutaneous SCC | 0.1
  New Primary Melanoma | 1.7
  GI Polyps | 0.03
  Pancreatitis | 0.2
  Potentiation of radiation toxicity | 1.4
  Prolongation of Cardiac Repolarization/ Arrhythmia | 17.0
  Other primary malignancy | 3.2
  Liver Injury | 14.1

4. Primary Outcome: Mean Cumulative Dose of Vemurafenib
Time Frame: Baseline up to end of treatment or death (maximum up to 46 months)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Grams | 501.283 (510.9121)

5. Primary Outcome: Duration of Vemurafenib Treatment
Description: Exposure excluding treatment interruptions: Duration during which participants actually took vemurafenib. Any time without dose-taken due to adverse events, non-compliance or any other reasons was not counted.
  Exposure including treatment interruptions: date of last dose - date of first dose + 1; duration during which participants actually took vemurafenib as well as duration on which medication was not taken were included in this calculation.
Time Frame: Baseline up to end of treatment or death (maximum upto 46 months)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Months
  Exposure excluding interruptions | 9.383 (9.6755) [0.03 to 11.24]
  Exposure including interruptions | 9.724 (9.9072)

6. Primary Outcome: Mean Total Vemurafenib Dose Per Day
Description: Exposure excluding treatment interruptions: Duration during which participants actually took vemurafenib. Any time without dose-taken due to adverse events, non-compliance or any other reasons was not counted.
  Exposure including treatment interruptions: date of last dose - date of first dose + 1; duration during which participants actually took vemurafenib as well as duration on which medication was not taken were included in this calculation. Average total dose per day: total actual dose taken divided by total actual days on treatment.
Time Frame: Baseline up to end of treatment or death (maximum up to 46 months)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Grams
  Average Total Dose Per Day Excluding Interruptions | 1.802 (0.2314)
  Average Total Dose Per Day Including Interruptions | 1.732 (0.2874)

7. Primary Outcome: Dose Intensity of Vemurafenib
Description: Dose intensity was defined as (total actual doses taken/total planned doses) *100, where total planned doses = prescribed doses * planned days on treatment, where planned days on treatment were defined as the interval between date of first dose and date of last dose.
Time Frame: Baseline up to end of treatment or death (maximum upto 46 months)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of planned dose
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of planned dose | 90.21 (14.966)

8. Secondary Outcome: Percentage of Participants With Improvement in Eastern Cooperative Group (ECOG) Performance Status
Description: ECOG Performance Status was measured on-therapy assessed participant's performance status on 5 point scale: 0 = fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50% of waking hours [hrs]), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Percentage of participants who had at least one point improvement from baseline at any assessment visit as well as at last study visit was reported.
Time Frame: Baseline, Day 1 of each 28 day cycle up to end of treatment (up to 46 months)
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of Participants
  At Least 1 Point Improvement at Any Visit | 24.7
  At Least 1 Point Improvement at Last Visit | 9.9

9. Secondary Outcome: Percentage of Participants Who Received Any Concomitant Medications
Description: Concomitant medications were all medications taken during the study, including those started before but ongoing at first dose. No medications for Melanoma were included. Percentage of participants who received at least one concomitant medication was reported.
Time Frame: Baseline up to 46 months
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of Participants | 93.8 [3.9 to 4.5]

10. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of Confirmed Complete Response (CR) or Partial Response (PR), as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: BOR was assessed by the investigator according to RECIST v1.1. BOR was defined as having confirmed CR or PR. CR: disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to less than (<) 10 millimeter (mm) in short axis; PR: at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesion, and no new lesions.
  Confirmed responses were those that persisted on repeat imaging greater than or equal to (>=) 4 weeks after initial response.
Time Frame: Baseline until first documentation of confirmed CR or PR (assessed at baseline, at Weeks 8, 16, as per institution standard of care thereafter but a minimum every 16 weeks thereafter until the end of the study [up to 46 months])
Population: Safety population. Number of participants analyzed = participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 2982
Percentage of Participants | 33.4 [31.7 to 35.1]

11. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time between the date of first confirmed CR or PR and date of first progression of disease (PD), or death, from any cause. Responses were assessed as per RECIST v1.1. CR: disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to < 10 mm in short axis; PR: at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesion, and no new lesions. Confirmed responses were those that persisted on repeat imaging >= 4 weeks after initial response. PD: at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesion.
Time Frame: From 1st documentation of confirmed CR or PR to PD or death, whichever occurred first (assessed at baseline, at Weeks 8, 16, as per institution standard of care thereafter but a minimum every 16 weeks thereafter until end of the study [up to 46 months])
Population: Safety population. Number of participants analysed=participants who achieved CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 996
Months | 7.4 [7.1 to 8.3]

12. Secondary Outcome: Time to Response
Description: Time to response was defined as the time between the date of first treatment and date of first confirmed CR or PR (assessed as per RECIST v1.1). CR: disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to < 10 mm in short axis; PR: at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesion, and no new lesions. Confirmed responses were those that persisted on repeat imaging >= 4 weeks after initial response.
Time Frame: Baseline until first documentation of confirmed CR or PR, whichever occurred first (assessed at baseline, at Weeks 8, 16, as per institution standard of care thereafter but a minimum every 16 weeks thereafter until the end of the study [up to 46 months])
Population: Safety population. Number of participants analyzed = participants with measurable disease at baseline.
Measure: Median (Full Range); unit: Months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 2982
Months | 1.84 [0.8 to 26.7]

13. Secondary Outcome: Percentage of Participants With PD Assessed According to RECIST v1.1 or Death
Description: PD was assessed according to RECIST v1.1. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesion.
Time Frame: Baseline until PD or death, whichever occurred first (assessed at baseline, at Weeks 8, 16, as per institution standard of care thereafter but a minimum every 16 weeks thereafter until the end of the study [up to 46 months])
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of Participants | 87.3 [0.8 to 26.7]

14. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time between the date of the first treatment and the date of first progression or death from any cause. PD was assessed according to RECIST v1.1. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesion.
Time Frame: as for outcome 13
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Months | 5.6 [5.5 to 5.8]

15. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline until death (maximum up to 46 months)
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Percentage of participants | 63.8 [11.5 to 12.7]

16. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from the date of first treatment to the date of death, regardless of the cause of death.
Time Frame: Baseline until death (maximum up to 46 months)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 3219
Months | 12.1 [11.5 to 12.7]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days post end of treatment (maximum up to 46 months)
Arm/Group | Vemurafenib
Serious Adverse Events (participants affected / at risk) | 1114/3219
Other Adverse Events (participants affected / at risk) | 2956/3219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=3219)
Anaemia (Blood and lymphatic system disorders) | 22
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Eosinophilia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 10
Angina pectoris (Cardiac disorders) | 5
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 15
Atrial flutter (Cardiac disorders) | 4
Cardiac failure (Cardiac disorders) | 6
Coronary artery disease (Cardiac disorders) | 3
Left ventricular dysfunction (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 7
Pericardial effusion (Cardiac disorders) | 7
Pericardial haemorrhage (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 7
Tachycardia (Cardiac disorders) | 1
Torsade de pointes (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperadrenalism (Endocrine disorders) | 1
Neovascular age-related macular degeneration (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 3
Uveitis (Eye disorders) | 6
Vitreous haemorrhage (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 16
Diverticular perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Heamatemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 3
Inguinal hernia (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 3
Jejunal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 4
Pancreatitis acute (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 17
Chest pain (General disorders) | 3
Chills (General disorders) | 1
Chronic fatigue syndrome (General disorders) | 1
Death (General disorders) | 7
Device dislocation (General disorders) | 1
Drug interaction (General disorders) | 1
Fatigue (General disorders) | 6
General physical health deterioration (General disorders) | 9
Malaise (General disorders) | 2
Multi-organ disorder (General disorders) | 1
Multi-organ failure (General disorders) | 2
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Visceral pain (General disorders) | 1
Pyrexia (General disorders) | 32
Sudden cardiac death (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 4
Cholelithiasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 3
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Food allergy (Immune system disorders) | 1
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 5
Blastocystis infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 5
Clostridium difficile infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 9
Escherichia bacteraemia (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 4
Groin abscess (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 3
H1N1 influenza (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 7
Lung infection (Infections and infestations) | 6
Oesophageal candidiasis (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 2
Pharyngotonsillitis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 31
Postoperative wound infection (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 7
Salmonella sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Septic shock (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 11
Urosepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 3
Vulvitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 4
Wound infection staphylococcal (Infections and infestations) | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Over dose (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Radiation injury (Injury, poisoning and procedural complications) | 2
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 7
C-reactive protein increased (Investigations) | 1
Gamma glutamyltransferase increased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 1
Lipase increased (Investigations) | 1
Liver function test abnormal (Investigations) | 3
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 68
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 260
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 43
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 259
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 3
Cerebral haematoma (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 14
Cerebrovascular accident (Nervous system disorders) | 10
Cognitive disorder (Nervous system disorders) | 3
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 10
Facial paresis (Nervous system disorders) | 1
Generalised tonic clonic seizure (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 3
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Intracranial pressure increased (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 2
Ischaemic stroke (Nervous system disorders) | 2
Nervous system disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Completed suicide (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 5
Psychotic disorder (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 2
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Renal colic (Renal and urinary disorders) | 2
Urinary tract disorder (Renal and urinary disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Acanthosis (Skin and subcutaneous tissue disorders) | 4
Actinic keratosis (Skin and subcutaneous tissue disorders) | 9
Angioedema (Skin and subcutaneous tissue disorders) | 2
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 3
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 3
Intermittent claudication (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 2
Hearnig impaired (Ear and labyrinth disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 3
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 3
Cataract (Eye disorders) | 2
Glaucoma (Eye disorders) | 2
Macular oedema (Eye disorders) | 2
Papilloedema (Eye disorders) | 2
Retinal artery occlusion (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Retinopathy (Eye disorders) | 1
Iritis (Eye disorders) | 2
Anal fistula (Gastrointestinal disorders) | 2
Anal skin tags (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteroocolitis (Gastrointestinal disorders) | 1
Faeces pale (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Leukoplakia oral (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertensive Crisis (Vascular disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 2
Asthenia (General disorders) | 2
Generalised oedema (General disorders) | 1
Impaired healing (General disorders) | 1
Surgical failure (General disorders) | 1
Euthanasia (General disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Hepatic failure (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 2
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1
Adnexal torsion (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Peyronie's disease (Reproductive system and breast disorders) | 1
Uterine cervical erosion (Reproductive system and breast disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 8
Nephrolithiasis (Renal and urinary disorders) | 1
Nephropathy (Renal and urinary disorders) | 1
Nephhropathy toxic (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Urinary fistula (Renal and urinary disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 3
Mania (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 2
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Blood glucose increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 3
Cystitis radiation (Injury, poisoning and procedural complications) | 1
Facial bone fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 4
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2
Acinetobacter infection (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Brain Abscess (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Cholecystitis infective (Infections and infestations) | 1
Colonic abscess (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 2
Hypopyon (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Localised infection (Infections and infestations) | 2
Lymph gland infection (Infections and infestations) | 1
Ophthalmic herpes zoster (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Subdiaphragmatic abscess (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adrenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral disorder (Nervous system disorders) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Monoplegia (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 2
Polyneuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 12
Simple partial seizure (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 3
Status epilepticus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1
Clostridium colitis (Infections and infestations) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=3219)
Diarrhoea (Gastrointestinal disorders) | 584
Nausea (Gastrointestinal disorders) | 718
Vomiting (Gastrointestinal disorders) | 449
Fatigue (General disorders) | 834
Pyrexia (General disorders) | 363
Weight decreased (Investigations) | 414
Decreased appetite (Metabolism and nutrition disorders) | 482
Arthralgia (Musculoskeletal and connective tissue disorders) | 1357
Myalgia (Musculoskeletal and connective tissue disorders) | 308
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 621
Headache (Nervous system disorders) | 458
Alopecia (Skin and subcutaneous tissue disorders) | 873
Dry skin (Skin and subcutaneous tissue disorders) | 538
Erythema (Skin and subcutaneous tissue disorders) | 327
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 830
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 678
Pruritus (Skin and subcutaneous tissue disorders) | 320
Rash (Skin and subcutaneous tissue disorders) | 556
Abdominal Pain (Gastrointestinal disorders) | 170
Constipation (Gastrointestinal disorders) | 196
Anaemia (Blood and lymphatic system disorders) | 215
Asthenia (General disorders) | 382
Oedema Peripheral (General disorders) | 238
Electrocardiogram QT prolonged (Investigations) | 521
Conjunctivitis (Infections and infestations) | 170
Nasopharyngitis (Infections and infestations) | 171
Sunburn (Injury, poisoning and procedural complications) | 318
Back Pain (Musculoskeletal and connective tissue disorders) | 191
Muscloskeletal Pain (Musculoskeletal and connective tissue disorders) | 222
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 276
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 227
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 266
Dysgeusia (Nervous system disorders) | 191
Insomnia (Psychiatric disorders) | 163
Cough (Respiratory, thoracic and mediastinal disorders) | 191
Actinic keratosis (Skin and subcutaneous tissue disorders) | 246
Palmar plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 193
Rash erythematous (Skin and subcutaneous tissue disorders) | 195
Rash Maculo- Papular (Skin and subcutaneous tissue disorders) | 179
Hypertension (Vascular disorders) | 264

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.